CLINICAL TRIAL: NCT03374800
Title: Re-EValuating the Inhibition of Stress Erosions: Prophylaxis Against Gastrointestinal Bleeding in the Critically Ill (The REVISE) Trial
Brief Title: Re-EValuating the Inhibition of Stress Erosions (REVISE) Trial
Acronym: REVISE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Canadian Critical Care Trials Group (Other); Australian and New Zealand Intensive Care Society Clinical Trials Group (Network); National Health and Medical Research Council, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CCT38473
Record Dates: First submitted 2017-11-21; First posted 2017-12-15 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Gastrointestinal Hemorrhage (Clinically Important, Upper)
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Sodium Chloride; Saline Solution; Pantoprazole

STUDY DESIGN:
Intervention Model Description: A prospective, international, multicentre, parallel group, concealed, blinded, randomized trial in critically ill invasively mechanically ventilated adults
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: blinded study drug and placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (0.9% saline) (Placebo Comparator): Withholding Stress ulcer prophylaxis (intravenous 0.9% saline as placebo)
  Interventions: Drug: Placebo (0.9% saline)
- Stress Ulcer Prophylaxis (Pantoprazole) (Active Comparator): pantoprazole 40mg powder for injection reconstituted with 0.9% saline
  Interventions: Drug: Pantoprazole

INTERVENTIONS:
Drug: Placebo (0.9% saline) — normal saline
  Other Names: normal saline; NaCl 0.9%
  Arms: Placebo (0.9% saline)
Drug: Pantoprazole — 40 mg powder for injection reconstituted with 0.9% saline
  Other Names: Protonix
  Arms: Stress Ulcer Prophylaxis (Pantoprazole)

SUMMARY:
Patients who are critically ill in the in the Intensive Care Unit (ICU), especially those who need a breathing machine, can develop ulcers in the stomach that bleed. To prevent bleeding, many such patients around the world receive a drug called pantoprazole that decreases acid production. However, today, compared to decades ago, critically ill patients rarely develop upper gastrointestinal bleeding. This decrease is likely due to modern medicine, better resuscitation and earlier feeding. There may also be harms associated with pantoprazole and other drugs that reduce acid levels in the stomach including lung infections (pneumonia) and bowel infections (Clostridioides difficile). Studies in this area are old and of modest quality. Therefore, it is difficult to know whether pantoprazole does decrease stomach bleeding these days, or whether the possible harms of lung and bowel infections are actually more common and more serious problems. The goal of this international study is to determine if, in critically ill patients using breathing machines, the use of pantoprazole is effective in preventing bleeding from stomach ulcers or whether it causes more problems such as lung infection (pneumonia) and bowel infection (Clostridioides difficile), or whether pantoprazole has no effect at all. Whether the harms are worth the benefits, and whether the benefits are worth the costs, will be determined by an economic analysis to inform patients, families, clinicians, and healthcare systems globally.

DETAILED DESCRIPTION:
Background: For 40 years, pharmacologic prevention of stress ulcer-related gastrointestinal (GI) bleeding with acid suppression has been the standard of care for invasively mechanically ventilated ICU patients. Worldwide, proton pump inhibitors (PPIs) are more commonly used than histamine-2-receptor antagonists. Observational studies and the latest network meta-analysis suggest that PPIs increase the risk of ventilator-associated pneumonia (VAP) and Clostridioides difficile infection (CDI). However, a recent large randomized trial showed that pantoprazole had no impact on the primary outcome of 90-day mortality. The secondary outcome (a composite of pneumonia, gastrointestinal bleeding, CDI and acute myocardial ischemia) was not different between the groups. Although pantoprazole was associated with a significantly lower rate of clinically important upper GI bleeding, some bleeding events required no blood transfusion, endoscopy or other diagnostic or therapeutic interventions, calling into question whether these bleeding events were truly patient-important. Further, patients with high illness severity on pantoprazole had a significant, unexplainable higher risk of death than those receiving placebo.

REVISE Pilot Trial: We completed the 91-patient REVISE Pilot Trial in Canada, Australia and Saudi Arabia, demonstrating a high consent rate (77.8%); recruitment rate (2.6 patients/month/center); and protocol adherence (96.8%), thereby successfully establishing the feasibility of a larger REVISE Trial.

Objectives of the REVISE Trial: To determine, among invasively mechanically ventilated patients, the effect of pantoprazole versus placebo on the primary efficacy outcome of clinically important upper GI bleeding, and the primary safety outcome of 90-day mortality. Secondary outcomes are VAP, CDI, acute kidney injury, ICU mortality, hospital mortality and patient-important upper GI bleeding. Tertiary outcomes are transfused packed red blood cells, serum creatinine, duration of mechanical ventilation, duration of ICU stay and duration of hospital stay.

Methods: We will include 4,800 ICU patients >18 years old who have an anticipated duration of mechanical ventilation of ≥48 hours. Exclusion criteria are acute or recent GI bleeding, dual antiplatelet therapy, combined antiplatelet and anticoagulant therapy, hopeless prognosis or intent to withdraw advanced life support, and previous enrolment in this or a confounding trial. Patients will be randomized in a fixed 1:1 allocation, stratified by center and pre-ICU acid suppression ('start or no start' strata, and 'continue or discontinue' strata). Research Coordinators will obtain informed consent using a deferred or a priori consent model. Study Pharmacists will obtain concealed allocation from the REVISE website; all research team and clinical team members, patients and families will be blinded. Patients will receive pantoprazole 40 mg or identical placebo intravenously daily while in ICU up to 90 days or until: 1) successful discontinuation of mechanical ventilation for >48 hours; 2) development of clinically important upper GI bleeding, or 3) death in ICU. Analyses will be by intention-to-treat with a sensitivity analysis restricted to patients receiving study drug on ≥ 80% of study days while mechanically ventilated per protocol.

Collaborations: REVISE will be conducted in collaboration with the Canadian Critical Care Trials Group, the Australian and New Zealand Critical Care Trials Group, other consortia and interested international investigators.

Ethical Imperative: Many factors converge to underscore the ethical imperative for REVISE. Critical care has evolved, research standards have improved, epidemiology may have changed, the risk:benefit and cost:benefit ratios of prophylaxis may have shifted. Thus, stress ulcer prophylaxis may need to be REVISED.

Relevance: Most invasively mechanically ventilated patients around the world receive daily stress ulcer prophylaxis, although variation exists such that some centers do not use any. Many RCTs of stress ulcer prophylaxis were conducted 10-30 years ago, several are at moderate or high risk of bias, and cointerventions may not reflect current critical care. A recent large trial raised concerns about death associated with pantoprazole in the most severely ill patient subgroup. Although clinically important upper GI bleeding events were less frequent, they may not have been patient-important, and there were no other benefits observed. Consensus in the scientific and clinical community is that equipoise remains regarding whether routine use of pantoprazole should continue for stress ulcer prophylaxis during critical illness. The question is especially important for patients who are receiving acid suppression pre-ICU, those who are receiving enteral nutrition, and those at high risk of death. Today, infectious complications of PPIs have emerged as potentially more common and serious than upper GI bleeding. The number needed to prophylax to prevent 1 GI bleed and the cost per GI bleed averted may be very high; furthermore, the number needed to harm to cause 1 episode of VAP or CDI may be low. Recent practice guidelines are conflicting. Remaining doubts about the effectiveness and safety of PPIs urge re-examination of universal prophylaxis for possible de-adoption. Aligned with the 'Choosing Wisely' Campaign, REVISE and the companion economic evaluation (E-REVISE) will be incorporated into guidelines to inform global practice.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or more.
2. Receiving invasive mechanical ventilation in an ICU and in the opinion of the treating ICU physician mechanical ventilation will not be discontinued before the end of the day after tomorrow.

Exclusion Criteria:

1. The treating clinician considers either Pantoprazole or placebo are indicated or contraindicated for this patient.
2. Pantoprazole contraindicated for patient due to local product information;

   Australia/New Zealand;
   * being treated with HIV protease inhibitors atazanavir or nelfinavir
   * being treated with high dose methotrexate (i.e., greater than 300 mg as part of a chemotherapy regimen).
   * documented cirrhosis or severe liver disease (for example as indicated by an INR greater than 5.0 due to underlying liver disease).

   Canada;
   * being treated with rilpivirine or atazanavir
   * patients who are hypersensitive to pantoprazole, substituted benzimidazoles, or to any ingredient in the formulation
3. Patients in whom a PPI or histamine 2 receptor antagonist (H2RA) is indicated due to active bleeding or increased bleeding risk, defined as patients with acute GI bleeding, severe oesophagitis or peptic ulcer disease within the previous 8 weeks, Zollinger Ellison syndrome, Barrett's oesophagus or any previous admission to hospital because of upper GI bleeding (patients receiving PPIs for mild dyspepsia or mild gastroesophageal reflux disease or an uncertain indication are not excluded).
4. Received invasive mechanical ventilation during this ICU admission for 72 hours or more.
5. Patients who have received more than 24 hours treatment (i.e., more than one daily dose equivalent) with a PPI or H2RA during this ICU admission.
6. Being treated with or need for dual anti-platelet therapy.
7. Admitted for palliative care or the ICU physician is not committed to continuing life-sustaining therapies at the time of enrolment.
8. Known or suspected pregnancy.
9. Physician, patient, or substitute decision maker (SDM) declines.
10. Previously enrolled in the REVISE trial
11. Enrolled in another trial for which co-enrolment is not approved.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4800 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Rate of clinically important upper gastro-intestinal bleeding | 90 days (In ICU or resulting in ICU readmission, censored at 90 days after randomization)
  Clinically important upper GI bleeding requires the presence of overt GI bleeding which is defined as one of the following;
  * Hematemesis
  * Overt nasogastric bleeding
  * Melena
  * Hematochezia
  PLUS (in the absence of another cause), at least one of the following in the 24 hours following overt GI bleeding:
  * Haemodynamic change defined as a spontaneous decrease in invasively monitored mean arterial pressure or non-invasive systolic or diastolic blood pressure of 20 mmHg or more or an orthostatic increase in pulse rate of 20 beats/minute and a decrease in systolic blood pressure of 10 mmHg, with or without vasopressor initiation, or increase
  * Vasopressor initiation
  * A decrease in haemoglobin of ≥ 20 g/l in a 24-hour period or less,
  * Transfusion of ≥2 units of packed red blood cells within 24 hours of bleeding to maintain stable haemoglobin or haemodynamics, or
  * Need for therapeutic intervention (e.g. angiography, surgery or endoscopic treatment of bleeding).
Primary Safety Outcome: 90 Day Mortality | 90 days post randomization
  Mortality status at day 90 post randomization

SECONDARY OUTCOMES:
Rate of ventilator associated pneumonia (VAP) in ICU | 90 Days (while in ICU,censored at 90 days after randomization)
  Diagnostic criteria for VAP include: previous mechanical ventilation for at least 48 hours, a new, progressive or persistent radiographic infiltrate on chest X-ray (without other obvious cause) plus at least 2 of the following 4 features:
  * fever or hypothermia (temperature >38 °C or <36 °C)
  * relative leukopenia or leukocytosis (WBC<4.0 or >12 x 10^9/L)
  * purulent sputum
  * gas exchange deterioration Using these uploaded data, the Clinical Pulmonary Infection Score is calculated. A score of 6 or greater is the primary definition of ventilator-associated pneumonia
Rate of Clostridioides difficile associated infection | 90 days (during the index hospital admission, censored at 90 days)
  We will use clinical features (diarrhea, ileus, toxic megacolon) and either microbiological evidence of toxin producing Clostridioides difficile or Pseudomembranous colitis on colonoscopy.
New initiation of treatment with renal replacement therapy in ICU | 90 Days (In the ICU, censored at 90 days)
  Rate of New initiation of treatment with renal replacement therapy in ICU
Rate of all-cause-in-hospital mortality | While in hospital, censored at 90 days after randomization
  hospital mortality
Rate of ICU mortality | While in the ICU, censored at 90 days after randomization
  ICU mortality
Rate of patient important upper GI bleeding in ICU or resulting in ICU readmission, censored at 90 days after randomization | Censored at 90 days after randomization
  Patient important upper GI bleeding in ICU or resulting in ICU readmission, censored at 90 days after randomization

OTHER OUTCOMES:
Total units of red blood cells transfused in the first 14 days of ICU stay | Censored at 14 days after randomization
  Total units of red blood cells transfused in the ICU in the first 14 days
Peak serum creatinine concentration in ICU | Censored at 90 days after randomisation
  Peak serum creatinine concentration in ICU
Duration of mechanical ventilation (days) | Censored at 90 days after randomisation
  Duration of mechanical ventilation (days)
ICU length of stay (days) | Censored at 90 days after randomisation
  ICU length of stay (days)
Hospital length of stay (days) | Censored at 90 days after randomisation
  Hospital length of stay (days)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Cook, MD, Principal Investigator — McMaster University
Locations (67):
- University of Nebraska - Nebraska Medical Center, Omaha, Nebraska, United States
- Australia (19):
  - Bankstown-Lidcombe Hospital, Bankstown, New South Wales
  - Blacktown Hospital, Blacktown, New South Wales
  - Sutherland Hospital, Caringbah, New South Wales
  - Gosford Hospital, Gosford, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Royal North Shore Hospital, Saint Leonards, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - Royal Brisbane Womens Hospital, Brisbane, Queensland
  - Ipswich Hospital, Ipswich, Queensland
  - Mater Hospital, South Brisbane, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Bendigo Health, Bendigo, Victoria
  - Geelong University Hospital, Geelong, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - Epworth Hospital, Melbourne, Victoria
- Brazil (2):
  - Sociedade Hospitalar Angelina Caron, Campina Grande do Sul
  - Beneficência Social Bom Samaritano, Governador Valadares
- Canada (41):
  - Foothills Hospital, Calgary, Alberta
  - Peter Lougheed Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Nanaimo Regional General Hospital, Nanaimo, British Columbia
  - Royal Columbian Hospital, New Westminster, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - Vancouver Island Health Authority, Victoria, British Columbia
  - St. Boniface Hospital, Winnipeg, Manitoba
  - Health Science Center Winnipeg, Winnipeg, Manitoba
  - Grace Hospital, Winnipeg, Manitoba
  - Saint John Regional Hospital, Saint John, New Brunswick
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - William Osler Hospital, McKenzie Health, Brampton Civic Hospital, Brampton, Ontario
  - Brantford General Hospital, Brantford, Ontario
  - Cambridge Memorial Hospital, Cambridge, Ontario
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Hamilton Health Science Center - General Hospital, Hamilton, Ontario
  - Hamilton Health Science Center - Juravinski Hospital, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - Grand River Hospital, Kitchener, Ontario
  - London Health Science Center (LHSC) - University Hospital, London, Ontario
  - London Health Science Center (LHSC) - Victoria Hospital, London, Ontario
  - North York General Hospital, North York, Ontario
  - Ottawa Health Research Institute - OHRI (General and Civic Hospital), Ottawa, Ontario
  - Niagara Health Services - St. Catharine's Hospital, St. Catharines, Ontario
  - Sunnybrook Health Science Center, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - University Health Network - Toronto Western Hospital, Toronto, Ontario
  - St. Joseph's Health Centre, Toronto, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Windsor Regional Hospital, Windsor, Ontario
  - Centre de recherche de l'Hôtel-Dieu de Lévis, Lévis, Quebec
  - Hôpital Maisonneuve Rosemont, Montreal, Quebec
  - Center Hospital University Montreal (CHUM), Montreal, Quebec
  - Centre Universitaire de Santé McGill / McGill University Health Centre, Montreal, Quebec
  - CIUSS du Nord de l'île de Montréal - Hôpital du Sacré-Cœur de Montréal, Montreal, Quebec
  - McGill University Health Centre - Montreal General Hospital, Montreal, Quebec
  - CHU de Québec-Université Laval - Hôpital Enfant-Jésus, Québec, Quebec
  - Institut Universitaire de cardiologie et de pneumologie de Québec Laval, Quebec, Québec, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
  - Regina General Hospital, Regina, Saskatchewan
- AL-Amiri Hospital, Kuwait City, Kuwait
- Maroof International Hospital, Islamabad, Pakistan
- King Abdulaziz Medical Center, Riyadh, Saudi Arabia
- Guys & St. Thomas Hospital, London, New Westminster, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Following the publication of REVISE, the dataset will be used for secondary observational studies addressing additional hypothesis-driven questions (e.g., predictors of gastrointestinal bleeding). Access by REVISE investigators will follow a submitted rationale, analysis plan and approval by the Management Committee. Requests for access to the dataset by external academic investigators will be considered following a submitted rationale, analysis plan and approval by the Management Committee and research ethics boards as relevant. Only de-identified data will be provided and will be transferred via a secure web portal. Requirements will be stipulated in a pre-specified data sharing agreement with investigators which aligns with each institution including the data sharing policy of The George Institute (https://www.georgeinstitute.org.au/data-sharing-policy.)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anticipated availability 2025 for up to 15 years.
Access Criteria: Following the publication of REVISE, the dataset will be used for secondary observational studies addressing additional hypothesis-driven questions (e.g., predictors of gastrointestinal bleeding). Access by REVISE investigators will follow a submitted rationale, analysis plan and approval by the Management Committee. Requests for access to the dataset by external academic investigators will be considered following a submitted rationale, analysis plan and approval by the Management Committee and research ethics boards as relevant. Only de-identified data will be provided and will be transferred via a secure web portal. Requirements will be stipulated in a pre-specified data sharing agreement with investigators which aligns with each institution including the data sharing policy of The George Institute (https://www.georgeinstitute.org.au/data-sharing-policy.)

REFERENCES:
- [Derived] Humphries B, Zytaruk N, Heels-Ansdell D, Lau V, Rochwerg B, Fowler R, Yao Y, Cook DJ, Xie F. Protocol for an economic evaluation alongside the Re-Evaluating the Inhibition of Stress Erosions (E-REVISE) trial. BMJ Open. 2025 Nov 9;15(11):e106841. doi: 10.1136/bmjopen-2025-106841. PMID 41213683
- [Derived] Clarke F, Hand L, Deane A, Zytaruk N, Hardie M, Arabi Y, Al-Fares A, Heels-Ansdell D, Dechert W, Ostermann M, Watpool I, Millen T, Muscedere J, English S, Boyd G, Sibley S, Peck L, Eastwood G, Duan E, Soth M, Freitag A, Vazquez-Grande G, Slessarev M, Ball I, Geagea A, Burns K, Binnie A, Mehta S, Tsang J, Burry L, D'Aragon F, Cook D. Coenrollment in a critical care trial: Characteristics and consequences. Contemp Clin Trials. 2025 Jul;154:107938. doi: 10.1016/j.cct.2025.107938. Epub 2025 May 14. PMID 40379131
- [Derived] Cook D, Deane A, Lauzier F, Zytaruk N, Guyatt G, Saunders L, Hardie M, Heels-Ansdell D, Alhazzani W, Marshall J, Muscedere J, Myburgh J, English S, Arabi YM, Ostermann M, Knowles S, Hammond N, Byrne KM, Chapman M, Venkatesh B, Young P, Rajbhandari D, Poole A, Al-Fares A, Reis G, Johnson D, Iqbal M, Hall R, Meade M, Hand L, Duan E, Clarke F, Dionne JC, Tsang JLY, Rochwerg B, Karachi T, Lamontagne F, D'Aragon F, St Arnaud C, Reeve B, Geagea A, Niven D, Vazquez-Grande G, Zarychanski R, Ovakim D, Wood G, Burns KEA, Goffi A, Wilcox ME, Henderson W, Forrest D, Fowler R, Adhikari NKJ, Ball I, Mele T, Binnie A, Trop S, Mehta S, Morgan I, Loubani O, Vanstone M, Fiest K, Charbonney E, Cavayas YA, Archambault P, Rewa OG, Lau V, Kristof AS, Khwaja K, Williamson D, Kanji S, Sy E, Dennis B, Reynolds S, Marquis F, Lellouche F, Rahman A, Hosek P, Barletta JF, Cirrone R, Tutschka M, Xie F, Billot L, Thabane L, Finfer S; REVISE Investigators. Stress Ulcer Prophylaxis during Invasive Mechanical Ventilation. N Engl J Med. 2024 Jul 4;391(1):9-20. doi: 10.1056/NEJMoa2404245. Epub 2024 Jun 14. PMID 38875111
- [Derived] Heels-Ansdell D, Billot L, Thabane L, Alhazzani W, Deane A, Guyatt G, Finfer S, Lauzier F, Myburgh J, Young P, Arabi Y, Marshall J, English S, Muscedere J, Ostermann M, Venkatesh B, Zytaruk N, Hardie M, Hammond N, Knowles S, Saunders L, Poole A, Al-Fares A, Xie F, Hall R, Cook D. REVISE: re-evaluating the inhibition of stress erosions in the ICU-statistical analysis plan for a randomized trial. Trials. 2023 Dec 6;24(1):796. doi: 10.1186/s13063-023-07794-z. PMID 38057875
- [Derived] Deane AM, Alhazzani W, Guyatt G, Finfer S, Marshall JC, Myburgh J, Zytaruk N, Hardie M, Saunders L, Knowles S, Lauzier F, Chapman MJ, English S, Muscedere J, Arabi Y, Ostermann M, Venkatesh B, Young P, Thabane L, Billot L, Heels-Ansdell D, Al-Fares AA, Hammond NE, Hall R, Rajbhandari D, Poole A, Johnson D, Iqbal M, Reis G, Xie F, Cook DJ; Canadian Critical Care Trials Group and the Australian and New Zealand Intensive Care Society Clinical Trials Group. REVISE: Re-Evaluating the Inhibition of Stress Erosions in the ICU: a randomised trial protocol. BMJ Open. 2023 Nov 15;13(11):e075588. doi: 10.1136/bmjopen-2023-075588. PMID 37968012
- [Derived] Dennis BB, Thabane L, Heels-Ansdell D, Dionne JC, Binnie A, Tsang J, Guyatt G, Ahmed A, Lauzier F, Deane A, Arabi Y, Marshall J, Zytaruk N, Saunders L, Finfer S, Myburgh J, Muscedere J, English S, Ostermann M, Hardie M, Knowles S, Cook D; REVISE Investigators the Canadian Critical Care Trials Group. Proton pump inhibitors in critically ill mechanically ventilated patients with COVID-19: protocol for a substudy of the Re-EValuating the Inhibition of Stress Erosions (REVISE) Trial. Trials. 2023 Aug 30;24(1):561. doi: 10.1186/s13063-023-07589-2. PMID 37644556

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-10): https://cdn.clinicaltrials.gov/large-docs/00/NCT03374800/Prot_SAP_000.pdf